CLINICAL TRIAL: NCT00506584
Title: A Randomized Study of Human Milk-Based Versus Bovine-based Nutrition for Very Low Birth Weight Pre-Term Infants
Brief Title: Randomized Study of Human-Milk Based Nutrition Versus Formula in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prolacta Bioscience (Industry)
Responsible Party: Martin L. Lee, PhD; Chief Scientific Officer, Prolacta Bioscience, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MPPF 001-2007
Record Dates: First submitted 2007-07-20; First posted 2007-07-25 (Estimated); Last update posted 2010-02-18 (Estimated); Status verified 2010-02

CONDITIONS: Infant, Very Low Birth Weight
Keywords: Human milk nutritional intervention; Pre-term, very low birth weight; Fortification of human breast milk
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Group 1, arm 1 (Experimental): Human breast milk + Prolact20/Neo20 (as needed) + Prolact+4 (initiated when nutrition volume reaches 100 mL/kg/day, where Prolact20/Neo 20 are donor human milk formulations at 20 cal/oz, Prolact+4 is a human-milk derived human milk fortified designed to add 4 cal/oz to 20 cal/oz human breast milk.
  Interventions: Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier
- Group1, Arm 2 (Experimental): Human breast milk + Prolact20/Neo20 (as needed) + Prolact+4 (initiated when nutrition volume reaches 40 mL/kg/day), where Prolact20/Neo 20 are donor human milk formulations at 20 cal/oz, Prolact+4 is a human-milk derived human milk fortified designed to add 4 cal/oz to 20 cal/oz human breast milk.
  Interventions: Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier
- Group 1, Arm 3 (Active Comparator): Human breast milk + bovine-based human milk fortifier (initiated when nutrition volume reaches 100 mL/kg/day) + pre-term formula (as needed)
  Interventions: Dietary Supplement: Human milk fortifier (bovine-based), pre-term formula
- Group 2, Arm 1 (Experimental): Prolact20/Neo20 + Prolact+4 (initiated when nutrition volume reaches 100 mL/kg/day), where Prolact20/Neo 20 are donor human milk formulations at 20 cal/oz, Prolact+4 is a human-milk derived human milk fortified designed to add 4 cal/oz to 20 cal/oz human breast milk.
  Interventions: Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier
- Group 2, Arm 2 (Active Comparator): Pre-term/term formula (minimum 20 cal/oz)
  Interventions: Dietary Supplement: Pre-term/term formula

INTERVENTIONS:
Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier — Human milk fortifier is initiated when nutrition volume reaches 100 mL/kg/day
  Other Names: Prolact20/Neo20; Prolact+4
  Arms: Group 1, arm 1
Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier — Human milk fortifier is initiated when nutrition volume reaches 40 mL/kg/day
  Other Names: Prolact20/Neo 20; Prolact+4
  Arms: Group1, Arm 2
Dietary Supplement: Human milk fortifier (bovine-based), pre-term formula — Bovine-based human milk fortifier is initiated when nutrition volume reaches 100 mL/kg/day
  Arms: Group 1, Arm 3
Dietary Supplement: Pasteurized human milk and pasteurized human milk fortifier — Human milk fortifier initiated when nutrition volume reaches 100 mL/kg/day
  Other Names: Prolact20/Neo20; Prolact+4
  Arms: Group 2, Arm 1
Dietary Supplement: Pre-term/term formula — Bovine milk-derived nutrition formulated for very low birth weight infants
  Arms: Group 2, Arm 2

SUMMARY:
The purpose of this study is to determine whether very low birth weight infants (less than or equal to 1250g or about 2 3/4 pounds) born prematurely fed a diet of only human milk and human milk-derived nutrition have better health outcomes than babies fed at least some formula (made from cow's milk)or formula-derived nutrition.

DETAILED DESCRIPTION:
The goal of this study is to evaluate the short-term effect (up to 90 days of life) of purely human-based nutrition using mother's own milk (when available), donor milk preparations and a human-based fortifier (Prolact+4) as needed when compared with mother's own milk supplemented with pre-term formula and using a bovine-based HMF (as needed for fortification of mother's own milk), i.e. "Study Group 1"; or, when mother's milk is not available, comparing the use of donor milk (plus human milk based fortification) with pre-term/term formula, i.e. "Study Group 2". In both instances the comparison will be based on the primary endpoint of days of TPN, and on parameters such as time to full enteral feeding (approximately 150-160 mL/kg/day), amount of IV fluid support, culture-proven sepsis, NEC, death, growth and short-term development, cultured-proven sepsis and incidence of feeding intolerance in either a 2-arm (human nutrition versus bovine nutrition: "Study Group 2") or 3-arm randomized design (human fortifier given when feedings reach 40 mL/kg/day, human fortifier given when feedings reach 100 mL/kg/day, and bovine-based HMF given when feedings reach 100 mL/kg/day [or pre-term formula if mother's milk is not available]: "Study Group 1").

Statistically, the study will attempt to evaluate a null hypothesis of equivalent results with respect to these parameters between either the three types of fortifications in "Study Group 1" or the two types of overall nutrition in "Study Group 2", as compared with an alternative of some inequality between the groups, i.e. letting μ be the mean number of days of TPN any of the study arms, then for "Study Group 1 the hypotheses may be written as:

H0: μ control = μ human 40 = μhuman 100 and HA: At least two of μ control, μ human 40, and μhuman 100 are not equal, where "control" is the bovine-based HMF group, "human 40" is the human fortifier group starting at 40 mL/kg/day (arm 2) and "human 100" is the human fortifier group starting at 100 mL/kg/day (arm 1). For "Study Group 2", the competing hypotheses are: H0: μ formula = μ human and HA: μ formula ≠ μ human , where "formula" is the pre-term/term formula group and "human" is the human-based (donor milk/human-based fortifier) group.

In addition, data will be collected on overall survival and length of stay in the NICU. Any baby that does not complete the full study period will be right-censored in this regard for the purposes of data evaluation. For centers that obtain long-term follow up (18-24 months) on their patients, data on developmental outcomes will be evaluated as available.

ELIGIBILITY:
Inclusion Criteria:

1. Birth weight between 500 and 1250g.
2. Have a reasonable expectation of survival for the maximum 90 day duration of the study.
3. In "Study Group 1", must be able to adhere to a feeding protocol involving mother's own milk and that may include donor human milk with fortification using a human-based product (Prolact+4) or fortification with a bovine-based human milk fortifier and the use of a pre-term/term formula; or in "Study Group 2" the use of donor human milk with Prolact+4 or a pre-term/term formula from the time that the infant initiates enteral feeding through day 90 of life, until discharge from the study institution, discharge home, death or the initiation of at least 50% total oral nutrition (4 complete feeds in a 24 hour period), whichever comes first.
4. Enteral feeding must begin before the 21st day of life.
5. Total parenteral nutrition (TPN) initiated within 48 hours after birth.
6. Informed consent obtained from parent or legal guardian.

Exclusion Criteria:

1. Less than a reasonable expectation of survival for the infant's particular gestational age through the study period (first 90 days of life, discharge to a non-study institution, discharge home, death or initiation of 50% oral nutrition, whichever comes first).
2. On any other clinical study affecting nutritional management during the study period.
3. Decision to not start minimum enteral feed before day 21 of life.
4. Decision to not start TPN within the first 48 hours after birth.
5. Unable to obtain informed consent from parent or legal guardian prior to the initiation of enteral feeding.
6. Presence of clinically significant congenital heart disease.
7. Presence of any major congenital malformations.
8. Reasonable potential for early transfer to a non-study institution.
9. Unable to participate for any reason based on the decision of the study investigator.

Ages: 1 Day to 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2007-07; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The primary measure of efficacy for the study is the number of days of TPN (total parenteral nutrition) | The first 90 days of life, discharge from the study institution or initiation of 50% oral nutrition (50% of the feeding volume in a given 24 hour period provided PO, or 4 complete PO feeds in a given 24 hour period), whichever comes first

SECONDARY OUTCOMES:
Weight gain and other measures of growth including length and head circumference | The first 90 days of life, transfer to non-study institution, or initiation of 50% oral feeding, whichever comes first
Daily amount of all nutrition | The first 90 days of life, transfer to non-study institution, or initiation of 50% oral feeding, whichever comes first
Time to discharge from the NICU and hospital | The first 90 days of life, transfer to non-study institution, or initiation of 50% oral feeding, whichever comes first
Frequency of occurrence of late-onset sepsis and necrotizing enterocolitis | The first 90 days of life, transfer to non-study institution, or initiation of 50% oral feeding, whichever comes first
Frequency of feeding intolerance | The first 90 days of life, transfer to non-study institution, or initiation of 50% oral feeding, whichever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Schanler, MD, Study Chair — Schneider Children's Hospital at North Shore
Locations (13):
- United States (12):
  - Alta Bates Summit Medical Center, Berkeley, California
  - University of California, San Diego Medical Center, San Diego, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Shands Children's Hospital, Gainesville, Florida
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Schneider Children's Hospital at North Shore, Manhasset, New York
  - Strong Memorial Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ben Taub Hospital/Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Utah Medical Center, Salt Lake City, Utah
- Innsbruck Children's Hospital, Innsbruck, Austria

REFERENCES:
- [Result] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Derived] Quigley M, Embleton ND, Meader N, McGuire W. Donor human milk for preventing necrotising enterocolitis in very preterm or very low-birthweight infants. Cochrane Database Syst Rev. 2024 Sep 6;9(9):CD002971. doi: 10.1002/14651858.CD002971.pub6. PMID 39239939
- [Derived] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Derived] Ghandehari H, Lee ML, Rechtman DJ; H2MF Study Group. An exclusive human milk-based diet in extremely premature infants reduces the probability of remaining on total parenteral nutrition: a reanalysis of the data. BMC Res Notes. 2012 Apr 25;5:188. doi: 10.1186/1756-0500-5-188. PMID 22534258